CLINICAL TRIAL: NCT05436093
Title: CLDN18.2 Targeting Nanobody Probe for PET Imaging in Solid Tumors
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Peking University Cancer Hospital & Institute (Other)
Responsible Party: Principal Investigator, Hua Zhu, Associate Professor, Peking University Cancer Hospital & Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 2022KT96
Record Dates: First submitted 2022-06-23; First posted 2022-06-28 (Actual); Last update posted 2024-01-25 (Actual); Status verified 2024-01

CONDITIONS: Solid Tumor
MeSH Terms: interventions — Fluorodeoxyglucose F18

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 68Ga-ACN376 (Experimental): Imaging cohort All study participants will be allocated to this arm (single-arm study). Study participants will undergo 68Ga-ACN376 PET/CT scan.
  Interventions: Drug: 18F-FDG

INTERVENTIONS:
Drug: 18F-FDG — All study participants will undergo one 18F-FDG PET/CT scan.

SUMMARY:
The objective of the study is to construct a noninvasive approach 68Ga-ACN376 PET/CT to detect the CLDN18.2 expression of tumor lesions in patients with Solid tumors and to identify patients benefiting from CLDN18.2 targeting treatment.

ELIGIBILITY:
Inclusion Criteria:

* 1. Aged >18 years old; ECOG 0 or 1;
* 2. Patients with solid tumors;
* 3. Has at least one measurable target lesion according to Response Evaluation Criteria in Solid Tumors (RECIST V1.1);
* 4. life expectancy >=12 weeks.

Exclusion Criteria:

* 1. Significant hepatic or renal dysfunction;
* 2. Is pregnant or ready to pregnant;
* 3. Cannot keep their states for half an hour;
* 4. Refusal to join the clinical study;
* 5. Suffering from claustrophobia or other mental diseases;
* 6. Any other situation that researchers think it is not suitable to participate in the experiment.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2022-06-23 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Standardized uptake value（SUV） | 2 years
  SUV is a semi-quantitative analysis index to describe the radioactive uptake of lesions, which has certain reference value for differentiating benign and malignant lesions。 The uptake of the tracer （68Ga-ACN376） in solid tumor lesions by measuring SUV on PET/CT.

CONTACTS AND LOCATIONS:
Overall Officials: Hua Zhu, Principal Investigator — Peking University Cancer Hospital & Institute
Locations (1):
- Beijing cancer hospital, Beijing, Beijing Municipality, China